CLINICAL TRIAL: NCT03043534
Title: The Impact of a Pre-Shave Gel and Brush in Males With Pseudofolliculitis Barbae
Brief Title: Pre-Shave Gel and Brush in Pseudofolliculitis Barbae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00034479
Record Dates: First submitted 2017-01-31; First posted 2017-02-06 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Pseudofolliculitis Barbae
MeSH Terms: conditions — pseudofolliculitis barbae | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gel and Brush (Experimental): The Experimental group of subjects will be given the study product Pre-Shave Gel and Brush. The gel and brush will be used prior to their normal shave routine. Subjects will shave at least 3 times weekly.
  Interventions: Other: shave gel; Other: Brush
- Control (No Intervention): Subjects will use their normal razors and shave products during the six week study. Subjects must shave at least 3 times weekly. No change in normal shaving is done in this group

INTERVENTIONS:
Other: shave gel — Non marketed pre-shave gel with the following INCI list of ingredients:
  WATER, GLYCERIN, DIMETHICONE, LAURETH-23, PETROLATUM, ACRYLAMIDE/SODIUM ACRYLOYLDIMETHYLTAURATE COPOLYMER, ISOPROPYL PALMITATE, HYDROXYETHYLCELLULOSE, FRAGRANCE, PEG-23M, C13-14 ISOPARAFFIN, DMDM HYDANTOIN, DISODIUM EDTA, LAURETH-7, IODOPROPYNYL BUTYLCARBAMATE
  Arms: Gel and Brush
Other: Brush — All subjects randomized to brush will use the brush with each shave
  Other Names: Oil of Olay cleansing brush
  Arms: Gel and Brush

SUMMARY:
This will be a randomized investigator blinded study of 40 men age 20-60 (inclusive) with symptoms of mild-moderate PFB based on Investigator Global Assessment (IGA). Subjects will be divided into two groups: the Control group of 20 subjects and the Experimental group of 20 Subjects. Subjects will be seen at Screening/Baseline, and 6 weeks.

All subjects will use their normal razors and shave products during the six week study. The Experimental group of subjects will also be given the study product Pre-Shave Gel and Cleansing Brush.

DETAILED DESCRIPTION:
This will be a randomized investigator blinded study of up to 40 men age 20-60 (inclusive) with symptoms of mild-moderate PFB based on Investigator Global Assessment (IGA). Subjects will be divided into two groups: the Control group of 20 subjects and the Experimental group of 20 Subjects. Subjects will be seen at Screening/Baseline, and 6 weeks.

All subjects will use their normal razors and shave products during the six week study. The Experimental group of subjects will also be given the study product Pre-Shave Gel and Cleansing Brush. The study gel and brush will be used prior to their normal shave routine.Quantitative lesion counts will be done by trained clinicians at each visit. Efficacy assessments include Investigator Global Assessment (IGA) scoring

ELIGIBILITY:
Inclusion Criteria:

1. Males with at least a two year history of the symptoms of PFB.
2. Must be age 20-60 years of age (inclusive).
3. Must wet shave using just a prep and blade razor at least 3 or more times per week, and be willing to continue that regimen during the study.
4. Must have Mild -to moderate PFB based on IGA rating scales. There are no lesion count inclusion requirements.

Exclusion Criteria:

1. Use of systemic (oral antibiotics) within the last 4 weeks.
2. Use of topical prescriptions (topical clindamycin, topical retinoids, topical metronidazole, topical sulfacetamide/sulfur, topical adapalene, benzoyl peroxide, salicylic acid, glycolic acid, retinol,chemical peels) or over-the-counter products the subject has used for PFB or Hair Growth within the last 2 weeks. Use of oral retinoids, laser therapy or electrolysis treatments or waxing in beard area in last 12 months.
3. Individuals who do not wet shave with a bladed razor, or who use electric shavers.
4. Subjects must not have used any type of cleansing or shave brush to the face for six weeks prior to Baseline.
5. Individuals who have removed a beard within last two months.
6. Individuals who have a history of alopecia areata of the face.
7. Confounding dermatological conditions that would, in the opinion of the principal investigator, preclude participation in this study such as:

   * Immune deficiency disease (HIV positive, AIDS, sarcoidosis)
   * On immunosuppressive drugs (e.g. oral corticosteroids)
   * Autoimmune disease (lupus, scleroderma, diabetes mellitus, vitiligo)
   * Koebnerizing diseases (e.g. psoriasis, lichens planus, (HPV) human papilloma virus, facial verruca, molluscum contagiosum)
   * Tuberculosis, Hepatitis B
   * History of Keloids
   * History of Herpes simplex in treated area
   * Bacterial infection of face including abscesses and draining sinuses of facial area
   * Cystic Acne, other acne in bearded area which interferes with shaving as well as the ability to distinguish PFB lesions from acne

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — les with psuedofolliculitis barbae
Enrollment: 29 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2016-10-12 (Actual); Study Completion 2016-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy McMIchael, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dept of Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gel and Brush | Control
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gel and Brush | Control | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 14 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Patient Global Severity Assessment- Mechanics of Shaving
Description: A total of the Patient's Global Assessment of mechanics of shaving based on following scale:
  How easy is it to… (please rank each phrase from 1 to 4; 1 = very easy, 2 = easy, 3 = difficult, 4 = very difficult)
  A) get a smooth shave after shaving? __________
  B) shave stubborn hairs? __________
  C) shave against the grain with little irritation? __________
  D) shave with the grain with little irritation? __________
  E) glide comfortably over your skin with the razor blade?
  For each subject, the total score could range from 5 -20, with lower numbers indicating better shave mechanics
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gel and Brush | Control
Number analyzed (Participants) | 15 | 14
score on a scale
  Baseline | 12.9 (2.6) | 12.4 (3.2)
  Week 6 | 8.5 (4.1) | 9.7 (4.8)

2. Secondary Outcome: Patient Global Severity Assessment (Degree of Itching, Burning and Stinging)
Description: Patient Global Severity Assessment measures itching/burning/stinging on the following scales:1 (no itching/no burning/no stinging at all) to 5 (very severe) the total score could range from 1-5 with the lower scores promoting a better outcome.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gel and Brush | Control
Number analyzed (Participants) | 15 | 14
score on a scale
  Baseline | 2.33 (1.04) | 2.64 (1.00)
  Week 6 | 1.46 (0.74) | 1.85 (0.94)

3. Secondary Outcome: Quality of Life Survey
Description: Quality of Life Survey will measure subjects' overall perception. For Shaving Experience, the total score could range from 6-42 with lower scores denoting better outcome measures.
  For Shaving Frustration, the total score could range from 3-21 with higher scores denoting better outcome measures.
  For Achieving Results, the total score could range from 3-21 with lower scores denoting better outcome measures.
  For Skin Feel, the total score could range from 3-21 with lower scores denoting better outcome measures.
  For Skin-Confidence, the total score could range from 4-28 with lower scores denoting better outcome measures.
  For Social Interactions, the total score could range from 6-42 with lower scores denoting better outcome measures.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gel and Brush | Control
Number analyzed (Participants) | 15 | 14
score on a scale
  Baseline Shaving Experience | 24.6 (10.3) | 23.5 (6.51)
  Baseline Shaving Frustrations | 13 (5.38) | 11.4 (2.59)
  Baseline Achieving Results | 12 (4.88) | 11.4 (4.55)
  Baseline Skin Feel | 13.2 (4.60) | 10.7 (4.59)
  Baseline Skin-Confidence | 16.3 (6.49) | 13.9 (5.2)
  Baseline Social Interactions | 19.4 (8.8) | 17.8 (5.6)
  Week 6 Shaving Experience | 12.5 (6.24) | 20.5 (6.5)
  Week 6 Shaving Frustrations | 14.6 (4.8) | 9.9 (2.9)
  Week 6 Achieving Results | 7.6 (5.1) | 8.0 (4.0)
  Week 6 Skin Feel | 6.5 (5.0) | 8.5 (4.6)
  Week 6 Self-Confidence | 10.8 (6.5) | 10.3 (5.2)
  Week 6 Social Interactions | 16.9 (10.4) | 13.3 (6.5)

4. Secondary Outcome: Lesions
Description: Lesions will be measured by counting papules, pustules, ingrown hairs, and Hyerpigmentation.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Gel and Brush | Control
Number analyzed (Participants) | 15 | 14
lesions
  Baseline | 23.7 (24.2) | 20.3 (2.1)
  Week 6 | 19.4 (18.5) | 16.1 (2.1)

5. Secondary Outcome: Investigator Global Assessment (IGA)
Description: Investigator Global Assessment (IGA) will measure disease severity using a scale 0 (Clear) - 5 (Very Severe) with the lower score grade denoting better outcome measures.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gel and Brush | Control
Number analyzed (Participants) | 15 | 14
units on a scale
  Baseline | 2.73 (0.79) | 2.57 (0.75)
  Week 6 | 2.06 (1.38) | 2.26 (0.85)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Gel and Brush | Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes